CLINICAL TRIAL: NCT02863913
Title: A Dose-escalation Phase I Trial of PD-1 Knockout Engineered T Cells for the Treatment of Muscle-invasive Bladder Cancer
Brief Title: PD-1 Knockout Engineered T Cells for Muscle-invasive Bladder Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Wujiang Liu, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11007965938
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2016-08

CONDITIONS: Invasive Bladder Cancer Stage IV
MeSH Terms: interventions — Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion. A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant). Patients will receive a total of 2, 3, 4 cycles of treatment.
  Interventions: Biological: PD-1 Knockout T Cells; Drug: Cyclophosphamide; Drug: IL-2
- Comparable group (Placebo Comparator): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will not be knocked out by CRISPR Cas9 in the laboratory (PD-1 Wild-type T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.
  Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant).
  Interventions: Drug: Cyclophosphamide; Drug: IL-2

INTERVENTIONS:
Biological: PD-1 Knockout T Cells — PD-1 Knockout T Cells and PD-1 wild-type T Cells will be made by Cell Biotech Co., Ltd. 2x107/kg T cells will be used for test group and comparable group separately.
  Arms: Test group
Drug: Cyclophosphamide — Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant).
  Other Names: cytophosphane
Drug: IL-2 — Interleukin-2 (IL-2) will be given in the following 5 days after cell infusion, 720000 international unit（IU）/Kg/day (if tolerant).
  Other Names: Interleukin-2 (IL-2)

SUMMARY:
This study will evaluate the safety of PD-1 knockout engineered T cells in treating metastatic advanced bladder cancer. Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a dose-escalation study of ex-vivo knocked-out, expanded, and selected PD-1 knockout-T cells from autologous origin. Patients are assigned to 1 of 3 treatment groups to determine the maximal tolerant dose. After the lower number of cycles are considered tolerant, an arm of the next higher number of cycles will be open to next patients. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified stage IV muscle-invasive bladder cancer with measurable lesions (On CT: longest diameter of tumoral lesion >=10 mm, shorted diameter of lymph node >=15 mm; measurable lesions should not have been irradiated)
* Progressed after all standard treatment
* Performance score: 0-1
* Expected life span: >= 6 months
* Toxicities from prior treatment has resolved. Washout period is 4 weeks for chemotherapy, and 2 weeks for targeted therapy
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Pathology is mixed type
* Emergent treatment of tumor emergency is needed
* Poor vasculature
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Compliance cannot be expected
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and tolerability of dose of PD-1 Knockout T cells using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients | Dose Escalation - Approximately 6 months

SECONDARY OUTCOMES:
Response Rate:Response will be evaluated according to RECIST v1.1 | 90 days
Progression free survival - PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to average 10 months
Overall Survival - OS | The time from randomization to death from any cause, assessed up to 2 years
Peripheral blood circulating tumor DNA | 6 weeks
  Peripheral circuiting tumor DNA is collected at baseline and 6 weeks after last treatment
Temporal Interleukin-2 change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interferon-γ change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interleukin-6 change in the peripheral blood | Baseline and 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
plan to share

REFERENCES:
- [Background] Bidnur S, Savdie R, Black PC. Inhibiting Immune Checkpoints for the Treatment of Bladder Cancer. Bladder Cancer. 2016 Jan 7;2(1):15-25. doi: 10.3233/BLC-150026. PMID 27376121
- [Background] Kim J. Immune checkpoint blockade therapy for bladder cancer treatment. Investig Clin Urol. 2016 Jun;57 Suppl 1(Suppl 1):S98-S105. doi: 10.4111/icu.2016.57.S1.S98. Epub 2016 May 26. PMID 27326412
- [Background] Aragon-Ching JB, Trump DL. Systemic therapy in muscle-invasive and metastatic bladder cancer: current trends and future promises. Future Oncol. 2016 Sep;12(17):2049-58. doi: 10.2217/fon-2016-0155. Epub 2016 Jun 16. PMID 27306417
- [Background] Festino L, Botti G, Lorigan P, Masucci GV, Hipp JD, Horak CE, Melero I, Ascierto PA. Cancer Treatment with Anti-PD-1/PD-L1 Agents: Is PD-L1 Expression a Biomarker for Patient Selection? Drugs. 2016 Jun;76(9):925-45. doi: 10.1007/s40265-016-0588-x. PMID 27229745
- [Background] Zibelman M, Plimack ER. Systemic therapy for bladder cancer finally comes into a new age. Future Oncol. 2016 Oct;12(19):2227-42. doi: 10.2217/fon-2016-0135. Epub 2016 Jul 12. PMID 27402371
- [Background] Donin NM, Lenis AT, Holden S, Drakaki A, Pantuck A, Belldegrun A, Chamie K. Immunotherapy for the Treatment of Urothelial Carcinoma. J Urol. 2017 Jan;197(1):14-22. doi: 10.1016/j.juro.2016.02.3005. Epub 2016 Jul 25. PMID 27460757
- [Derived] Yi L, Li J. CRISPR-Cas9 therapeutics in cancer: promising strategies and present challenges. Biochim Biophys Acta. 2016 Dec;1866(2):197-207. doi: 10.1016/j.bbcan.2016.09.002. Epub 2016 Sep 15. PMID 27641687